CLINICAL TRIAL: NCT05947331
Title: Graded Anderson Versus Kestenbaum Procedure for Correction of Head Turn in Idiopathic Infantile Nystagmus
Brief Title: Correction of Head Turn in Idiopathic Infantile Nystagmus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Sara Fawzy Ibrahim Mahmoud Eid, Assisstant lecturer of ophthalmology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Head Turn in nystagmus
Record Dates: First submitted 2023-07-05; First posted 2023-07-17 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Infantile Nystagmus Syndrome

STUDY DESIGN:
Intervention Model Description: The patients with infantilenystagmus related head turn are divided randomly in two groups according to the surgical procedure to be performed Group I (Graded Anderson procedure);Group II (Kestenbaum procedure)
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Graded Anderson procedure) (Active Comparator): patients with idiopathic infantile nystagmus related head turn corrected by graded Anderson procedure.
  Interventions: Procedure: Graded Anderson procedure
- Group II (Kestenbaum procedure) (Active Comparator): patients with idiopathic infantile nystagmus related head turn corrected by Kestenbaum procedure.
  Interventions: Procedure: Kestenbaum procedure

INTERVENTIONS:
Procedure: Graded Anderson procedure — In graded Anderson proceduren only recession of yoke muscles is done.
  Arms: Group I (Graded Anderson procedure)
Procedure: Kestenbaum procedure — In Kestenbaum procedure, recession of yoke muscles and resection of their antagonists is done based on Parks table for Kestenbaum procedure according to the preoperative amount of head turn.
  Arms: Group II (Kestenbaum procedure)

SUMMARY:
Infantile nystagmus is involuntary, bilateral, conjugate and rhythmic oscillations of the eyes which may present at birth or develop within the first 6 months of life. It may be idiopathic appearing without visual or neurological impairment or may be secondary to an afferent visual defect such as foveal hypoplasia, congenital cataract, retinal dystrophy or optic atrophy. Aiming at improving outcome of head turn in idiopathic infantile nystagmus, comparison between the efficacy and safety of graded Anderson procedure and Kestenbaum procedure is essential.

DETAILED DESCRIPTION:
Infantile nystagmus related abnormal head position is noted according to the axis, it can be anomalous horizontally (right or left head turn), vertically (chin up or down), torsionally (right or left head tilt) or in a mixed pattern. A head turn to right or left is the most common compensatory posture encountered in patients with infantile nystagmus with an eccentric null position. A prolonged head turn (HT) may interfere with the social interactions and the quality of life and may lead to skeletal deformities in the cervical spine with postural dysfunction and impaired movement pattern. Thus, the correction of an abnormal head turn is important to enlarge the visual field, to eliminate the possibility of abnormal contracture of the neck muscles and to permit an adequate vision.Various extraocular muscle surgeries have been advised to correct infantile nystagmus-related HT. Despite being the most common surgical technique used till today for correction of head turn related to nystagmus, Kestenbaum procedure has variable long- term results, limited success rate and involves four rectus muscles (recession/ resection). In graded Anderson procedure, only yoke muscle recession is done based on the amount of initial head turn leaving two untouched muscles.

ELIGIBILITY:
Inclusion Criteria:

Orthophoric Patients with idiopathic infantile nystagmus related head turn (≥20 degrees - ≤ 45 degrees) that is verified at least twice in two separate visits.

Exclusion Criteria:

1. Patients with infantile nystagmus secondary to ocular diseases
2. Patients with infantile nystagmus with associated strabismus.
3. Previous squint, scleral buckling or glaucoma surgeries.
4. Associated systemic or neurological disorders.
5. Patients with anisometropia ≥ 5D.
6. Patients with nystagmus attenuated at near

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Degree of head turn | Base line and 6 months postoperatively.
  assess the change from Baseline degree of head turn at 6 months postoperatively using protractor goniometer

SECONDARY OUTCOMES:
Best corrected visual Acuity | Base line and 6 months postoperatively
  assess the change from Baseline best corrected visual acuity at 6 months postoperatively
stereopsis | Base line and 6 months postoperatively.
  assess the change from Baseline stereopsis at 6 months postoperatively using titmus fly test
complications | 6 months postoperatively
  report intraoperative and postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Y EL-Mashad, Dr., Study Director — professor of ophthalmology, Zagazig University; Emad M El-Hady, Dr., Study Chair — professor of ophthalmology, Zagazig University; Mostafa A Abdel-Aziz, Dr., Study Chair — Assisstant professor of ophthalmology, Zagazig University; sara F Ibrahim Mahmoud Eid, Master, Principal Investigator — Assisstant lecturer of Ophthalmology, Zagazig University
Locations (1):
- Zagazig University, Zagazig, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
names and affiliations of the participants

REFERENCES:
- [Background] Abadi RV, Bjerre A. Motor and sensory characteristics of infantile nystagmus. Br J Ophthalmol. 2002 Oct;86(10):1152-60. doi: 10.1136/bjo.86.10.1152. PMID 12234898
- [Background] Hertle RW. Nystagmus in infancy and childhood: characteristics and evidence for treatment. Am Orthopt J. 2010;60:48-58. doi: 10.3368/aoj.60.1.48. PMID 21061884
- See also: Management of Congenital Nystagmus with and without Strabismus — https://rdcu.be/df8N8
- See also: Graded Anderson procedure for correcting abnormal head posture in infantile nystagmus — https://rdcu.be/df8Mh
- See also: High-dose Anderson operation for nystagmus-related anomalous head turn — https://rdcu.be/df8MT